CLINICAL TRIAL: NCT02308540
Title: A Phase 1/2, Prospective,Randomized, Active-Controlled, Double-Blind, Age De-escalation Study to Evaluate the Safety, Tolerability, Immunogenicity of Serum Institute of India's PCV10 in Healthy Adults, Toddlers, and Infants
Brief Title: Safety and Immunogenicity of a 10 Valent Pneumococcal Conjugate Vaccine (SIILPCV10) in Healthy Adults, Toddlers, Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-017
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Adult SIILPCV10 (Experimental): Single dose of SIILPCV10 on day 0
  Interventions: Biological: SIILPCV10
- Adult Pneumovax 23 (Active Comparator): Single dose of Pneumovax 23 on day 0
  Interventions: Biological: Pneumovax 23
- Toddler SIILPCV10 (Experimental): Single dose of SIILPCV10 on day 0
  Interventions: Biological: SIILPCV10
- Toddler Prevenar 13 (Active Comparator): Single dose of Prevenar 13 on day 0
  Interventions: Biological: Prevenar 13
- Infants SIIL PCV10 (Experimental): A three-dose series of SIILPCV10 on day 0, day 28, and day 56
  Interventions: Biological: SIILPCV10
- Infants Prevenar 13 (Active Comparator): A three-dose series of Prevenar 13 on day 0, day 28, and day 56
  Interventions: Biological: Prevenar 13
- Infant Booster Dose SIILPCV 10 (Experimental): One dose of SIILPCV 10 at 9 months of age
  Interventions: Biological: SIILPCV10
- Infant Booster Dose Prevenar 13 (Active Comparator): One dose of SIILPCV 10 at 9 months of age
  Interventions: Biological: Prevenar 13

INTERVENTIONS:
Biological: SIILPCV10 — 10-valent Pneumococcal Conjugate Vaccine (SIILPCV10) at a dosage of 2 µg for each serotype polysaccharide, except 4 µg for 6B serotype, conjugated to a carrier protein (CRM197), with adjuvant (aluminum phosphate [alum]) and preservative (thiomersal).
  Arms: Adult SIILPCV10; Infant Booster Dose SIILPCV 10; Infants SIIL PCV10; Toddler SIILPCV10
Biological: Pneumovax 23 — 23-valent Pneumococcal Polysaccharide Vaccine (Pneumovax 23; MSD Pharmaceuticals) for the adult cohort.
  Other Names: 23-valent Pneumococcal Polysaccharide Vaccine
  Arms: Adult Pneumovax 23
Biological: Prevenar 13 — 13-valent Pneumococcal Conjugate Vaccine (Prevenar 13; Pfizer-Wyeth) for the toddler and infant cohorts
  Other Names: 13-valent Pneumococcal Conjugate Vaccine
  Arms: Infant Booster Dose Prevenar 13; Infants Prevenar 13; Toddler Prevenar 13

SUMMARY:
Phase 1/2, Prospective, Single Center, Randomized, ActiveControlled, Double-Blind, Age De-escalation Study to assess the safety and tolerability of SIILPCV10 administered as a single-dose regimen to healthy Gambian pneumococcal conjugate vaccine (PCV)-naïve young adults and PCV-primed toddlers through 4 weeks post vaccination.

Each adult and toddler subject will undergo a total of 4 clinic visits. Each infant subject will undergo a total of 9 scheduled visits. Blood will be collected from all subjects during the screening visit for safety and potential immunological assessments, and 28 days after completion of the vaccination schedule for immunological assessments. For adults, the vaccine was given intramuscularly into the mid-deltoid muscle of nondominant arm using a 24-gauge needle. For toddlers and infants, the vaccine will be given IM into the anterolateral aspect of the left thigh. Blood will be collected from adults and toddlers for safety labs at the Day 7 post-vaccination visit.

DETAILED DESCRIPTION:
This was a prospective, single-center, randomized, active-controlled, double-blind, age de escalation study in healthy Gambian PCV-naïve adults (18-40 years old), PCV primed toddlers (12-15 months old) and PCV-naïve infants (6-8 weeks old).

In the adult cohort, at least 34 eligible PCV-naïve adults (18-40 years old) were planned to be randomized into the study to receive a single dose of either SIILPCV10 or Pneumovax 23 in a 1:1 ratio on Day 0 (V1), with stratification by sex (although no fixed proportion of males and females was required in the cohort as a whole).

In the toddler cohort, at least 112 eligible PCV-primed toddlers (12-15 months old) were planned to be randomized into the study to receive a single dose of either SIILPCV10 or Prevenar 13 in a 1:1 ratio on Day 0 (V1).

Each adult and toddler subject underwent a total of 4 clinic visits, including at least 1 screening visit (V0) no more than 14 days prior to Day 0, a vaccination visit on Day 0 (V1), and follow-up clinic visits at 7 (+3) and 28 (+14) days after vaccination (V2 and V3, respectively). A total of 3 blood samples were obtained for laboratory safety and immunogenicity assessments.

In the infant cohort, at least 200 eligible PCV-naïve infants (6 to 8 weeks old) were randomized into the study to receive 3 doses of either SIILPCV10 or Prevenar 13 in a 1:1 ratio along with standard Expanded Program on Immunisation (EPI) vaccinations (pentavalent diphtheria, tetanus, whole-cell pertussis, hepatitis B, and Haemophilus influenzae type b combined vaccine [DTwP-HepB-Hib], oral poliovirus vaccine [OPV], rotavirus vaccine [RV], and inactivated poliovirus vaccine [IPV]).

Each infant subject underwent a total of 9 scheduled visits for the primary series: at least 1 screening visit (V0); 3 primary vaccination visits at 28 (+14)-day intervals (V1, 3, 5); follow-up clinic visits at 7 (+3) days after each primary vaccination (V2, 4, 6); and 2 follow-up visits 28 and 84 days after the last primary vaccination (V7 and V8, respectively). Windows for follow-up and subsequent vaccination visits were calculated based on the actual calendar date of the prior vaccination, rather than relative to the day of randomization. Vaccinations included the blinded PCV study vaccine (SIILPCV10 or Prevenar 13) and the unblinded EPI vaccines (DTwP-HepB-Hib, OPV, RV, and IPV).

A total of 2 blood samples were obtained for the primary series (V0 and V7), with the first sample used for safety laboratory eligibility assessment, and if randomized, for baseline immunogenicity testing. Immunogenicity testing was also done on the second sample.

During the supplemental booster phase, infant subjects underwent 2 additional visits: a fourth (booster) vaccination visit (V9) at ≥ 9 months of age, and a follow-up visit 28 days after the booster dose (V10). The EPI vaccines scheduled for 9 months of age in The Gambia were not given as part of the study. However, study personnel contacted parents of infant subjects to remind them of the need to attend this EPI vaccination visit at the due date to allow for effective scheduling of the subsequent booster. The vaccine (SIILPCV10 or Prevenar 13) was given at least 4 weeks after the routine EPI vaccines given at 9 months of age in The Gambia (measles and rubella, yellow fever, and OPV). Infants who received SIILPCV10 at V9 were offered a booster dose of Prevenar 13 at least 56 days following the SIILPCV10 boost. Immunogenicity testing was performed on 2 additional blood samples collected during the booster phase (V9 and V10).

In the adult and toddler cohorts, on the day of vaccination, a malaria rapid test was performed using a finger prick to rule out parasitemia and a urine pregnancy test was performed (in adult women who were not surgically sterile) to rule out pregnancy before final eligibility was confirmed and randomization occurred. In the infant cohort, on each day of vaccination, a malaria rapid test was performed using a finger prick to rule out parasitemia before vaccination occurred. Any infant showing signs of acute illness or abnormal vital signs on the day of vaccination were not vaccinated until recovery was documented by the study team.

After all vaccinations, subjects were monitored for solicited reactogenicity. All adult and toddler subjects were monitored for AEs at each clinic visit until V3, and ongoing AEs at study exit were followed until last subject last visit (LSLV). Infant subjects were monitored for AEs at each clinic visit until V8. For infants who participated in the booster phase of the study, AEs were recorded at V10, and any conditions present at V9 were considered baseline.

SAS software was used to analyze data.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy adults (18-40 yrs), toddlers (12-15 mo), full term infants (6-8 wks) and ≥ 3.5 kg

  * Able to provide informed consent (for themselves or child)
  * Willing to comply with study requirements and procedures.
  * Toddlers have completed their Gambian infant EPI schedule
  * Infants who have received the birth doses of BCG, HepB and OPV but who have not received any additional vaccines.
  * Infants and toddlers with a weight-to-height Z score of ≥ -2.
  * Subjects resident in the study area with no plans to travel outside the study area during the period of study participation.

Exclusion Criteria:

* Use of any investigational medicinal product within 90 days prior to randomization and throughout the study.
* Ingestion of herbal or other traditional local medication within 14 days of randomization.
* Adults and infants who have previously been vaccinated against S. pneumoniae.
* History of S. pneumoniae infection confirmed by culture from a normally sterile site.
* History of allergic disease or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the study vaccines.
* History of anaphylactic shock.
* Screening laboratory test or vital signs outside the normal range.
* HIV-positive or HbsAg- positive based on testing during screening.
* Acute illness (moderate or severe) and/or fever (axillary temperature of ≥ 38.0°C for adults or ≥ 37.5°C for toddlers and infants).
* Use of antibiotics within 5 days of randomization (excluding treatment for malaria).
* A positive test for malaria at time of screening, which remains positive post treatment when retested at time of randomization (Day 0).
* Administration of any non-study vaccine within 30 days prior to administration of study vaccine or planned vaccination during the course of study participation.
* Chronic administration of immunosuppressant or other immune modifying drugs prior to the administration of the study. The use of topical and inhaled glucocorticoids will be permitted.
* Administration of immunoglobulins and/or any blood products within the 6 months prior to administration of the study vaccine or during the study period.
* History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding.
* Employee of, or direct descendant of any person employed by the Sponsor, the CRO, the PI, study site personnel, or site.

Adults only

* Recent history or signs of alcohol or substance abuse.
* History of major psychiatric disorder.
* Female adult subjects who are pregnant or breast-feeding. Infants/Toddlers only
* Family history of suspected primary immunodeficiency in first-degree relative.
* Had a sibling die suddenly and without apparent other cause or preceding illness in the first year of life.
* Evidence of a clinically significant congenital abnormality as judged by the PI.
* Evidence of fetal alcohol syndrome or maternal history of alcohol abuse during pregnancy.
* History of meningitis, seizures or any neurological disorder.
* Evidence of exposure to an HIV-positive individual through maternal fetal transmission, breast milk, or other bloodborne mechanisms

Ages: 4 Weeks to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 346 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, MD PhD, Principal Investigator — Medical Research Council (MRC) Unit, The Gambia
Locations (1):
- Medical Research Council (MRC) Unit, The Gambia, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clarke E, Bashorun AO, Okoye M, Umesi A, Badjie Hydara M, Adigweme I, Dhere R, Sethna V, Kampmann B, Goldblatt D, Tate A, Weiner DH, Flores J, Alderson MR, Lamola S. Safety and immunogenicity of a novel 10-valent pneumococcal conjugate vaccine candidate in adults, toddlers, and infants in The Gambia-Results of a phase 1/2 randomized, double-blinded, controlled trial. Vaccine. 2020 Jan 10;38(2):399-410. doi: 10.1016/j.vaccine.2019.08.072. Epub 2019 Dec 14. PMID 31843266

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adult cohort: 43 screened and 9 screen failures Toddler cohort: 173 screened and 61 screen failures Infant cohort: 262 screened and 62 screen failures
Groups:
- Infants SIILPCV10: A three-dose series of SIILPCV10 on day 0, day 28, and day 56; Booster dose of SIILPCV 10 at 9 months of age.
  SIILPCV10: 10-valent Pneumococcal Conjugate Vaccine (SIILPCV10) at a dosage of 2 µg for each serotype polysaccharide, except 4 µg for 6B serotype, conjugated to a carrier protein (CRM197), with adjuvant (aluminum phosphate [alum]) and preservative (thiomersal).
Period: Overall Study
Arm/Group | Adult SIILPCV10 | Adult Pneumovax 23 | Toddler SIILPCV10 | Toddler Prevenar 13 | Infants SIILPCV10 | Infants Prevenar 13
Started | 17 | 17 | 56 | 56 | 100 | 100
Randomized | 17 | 17 | 56 | 56 | 100 | 100
Vaccinated | 17 | 17 | 56 | 56 | 100 | 100
Completed | 17 | 17 | 56 | 56 | 100 | 99
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Adults--PCV 10; Toddler--PCV 10: Single dose of SIILPCV 10 on Day 0
- Adults--Pneumovax 23: Single dose of Pneumovax 23 on Day 0
- Toddler--Prevenar 13: Single dose of Prevenar 13 on Day 0
- Infant--PCV 10: A 3-dose series of SIILPCV 10 on Day 0, Day 28, and Day 56.
- Infant--Prevenar 13: A 3-dose series of Prevenar 13 on Day 0, Day 28, and Day 56.
- Infant Boost--PCV 10: [Subset of infants in main study] Booster dose of SIILPCV 10 at 9 months of age
- Infant Boost--Prevenar 13: [Subset of infants in main study] Booster dose of Prevenar 13 at 9 months of age
- Total: Total of all reporting groups
Arm/Group | Adults--PCV 10 | Adults--Pneumovax 23 | Toddler--PCV 10 | Toddler--Prevenar 13 | Infant--PCV 10 | Infant--Prevenar 13 | Infant Boost--PCV 10 | Infant Boost--Prevenar 13 | Total
Number analyzed (Participants) | 17 | 17 | 56 | 56 | 100 | 100 | 49 | 47 | 442
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only adults are included in this category. Infants and toddlers are included in their own separate categories.
  years
    Adults in years: number analyzed (Participants) | 17 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 34
    Adults in years | 25.9 (4.1) | 25.9 (4.4) |  |  |  |  |  |  | 25.9 (4.1)
Age, Continuous [Mean (Standard Deviation); unit: Days] — Population: Only infants are represented here. Adults, toddlers and infants in booster cohort are represented separately.
  Days
    Infants--Age in Days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 100 | 0 | 0 | 200
    Infants--Age in Days |  |  |  |  | 47.2 (4) | 47.3 (3.8) |  |  | 47.2 (3.9)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Only toddlers are represented here. Adults and infants are presented separately.
  Months
    Toddler--Age in months: number analyzed (Participants) | 0 | 0 | 56 | 56 | 0 | 0 | 0 | 0 | 112
    Toddler--Age in months |  |  | 13.3 (0.9) | 13.3 (0.8) |  |  |  |  | 13.3 (0.9)
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: This includes data from infant booster cohort. Data from adults, toddlers and infants are represented separately
  months
    Infant Booster age in Months: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 47 | 96
    Infant Booster age in Months |  |  |  |  |  |  | 11.4 (0.8) | 11.5 (0.9) | 11.4 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 30 | 32 | 52 | 49 | 20 | 20 | 211
  Male | 13 | 13 | 26 | 24 | 48 | 51 | 29 | 27 | 231
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 17 | 17 | 56 | 56 | 100 | 99 | 49 | 47 | 441
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Gambia | 17 | 17 | 56 | 56 | 100 | 100 | 49 | 47 | 442
Ethnicity [Count of Participants; unit: Participants]
  Mandinka | 10 | 7 | 28 | 27 | 42 | 55 | 23 | 28 | 220
  Wolof | 3 | 1 | 4 | 11 | 18 | 10 | 9 | 2 | 58
  Fula | 2 | 4 | 6 | 7 | 12 | 10 | 6 | 5 | 52
  Jola | 1 | 2 | 11 | 3 | 12 | 12 | 5 | 3 | 49
  Serahule | 0 | 2 | 2 | 2 | 5 | 3 | 1 | 3 | 18
  Serere | 0 | 0 | 3 | 3 | 8 | 5 | 5 | 5 | 29
  Manjago | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  Other | 1 | 0 | 1 | 3 | 3 | 4 | 0 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Adult and Toddler Subjects Experiencing Local and Systemic Reactogenicity, by Severity
Description: Local and systemic reactogenicity of the study vaccine was evaluated for severity by toxicity grading scale (0 [none], 1 [mild], 2 [moderate], 3 [severe], 4 [potentially life threatening]) and relatedness to the vaccination. Injection site events were by definition considered related to study vaccine. Reactogenicity was monitored at the following times:
  * At 60 (± 15) minutes following primary vaccination
  * Daily by field workers during Days 1 to 6 post vaccination
  * In the clinic on Day 7 (+3) following each vaccination (Visit 2 for adults and toddlers).
Time Frame: 7 days
Population: All subjects who received at least 1 study vaccination and had at least 1 post vaccination safety measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Adults--PCV10: A single dose of SIILPCV 10 at Day 0
- Adults--Pneumovax 23: A single dose of Pneumovax 23 at Day 0
- Toddler--PCV 10: A single dose of SIIL PCV 10 at Day 0
- Toddler--Prevenar 13: A single dose of Prevenar 13 at Day 0
Arm/Group | Adults--PCV10 | Adults--Pneumovax 23 | Toddler--PCV 10 | Toddler--Prevenar 13
Number analyzed (Participants) | 17 | 17 | 56 | 56
Participants
  Temperature above 37.5 C: Grade 1 | 0 | 0 | 5 | 6
  Temperature above 37.5 C: Grade 2 | 0 | 0 | 2 | 4
  Temperature above 37.5 C: Grade 3 | 0 | 0 | 2 | 1
  Temperature above 37.5 C: Grade 4 | 0 | 0 | 0 | 0
  Temperature above 37.5 C: None reported/normal (temp) | 17 | 17 | 47 | 45
  Rash: Grade 1 | 0 | 0 | 1 | 0
  Rash: Grade 2 | 0 | 0 | 1 | 0
  Rash: Grade 3 | 0 | 0 | 0 | 0
  Rash: Grade 4 | 0 | 0 | 0 | 0
  Rash: None reported/normal (temp) | 17 | 17 | 54 | 56
  Fatigue/Malaise/Drowsiness (inf/tod): Grade 1 | 1 | 2 | 5 | 0
  Fatigue/Malaise/Drowsiness (inf/tod): Grade 2 | 0 | 0 | 1 | 0
  Fatigue/Malaise/Drowsiness (inf/tod): Grade 3 | 0 | 0 | 0 | 0
  Fatigue/Malaise/Drowsiness (inf/tod): Grade 4 | 0 | 0 | 0 | 0
  Fatigue/Malaise/Drowsiness (inf/tod): None reported/normal (temp) | 16 | 15 | 50 | 56
  Myalgia/Arthralgia (adults only): Grade 1 | 0 | 0 | 0 | 0
  Myalgia/Arthralgia (adults only): Grade 2 | 0 | 0 | 0 | 0
  Myalgia/Arthralgia (adults only): Grade 3 | 0 | 0 | 0 | 0
  Myalgia/Arthralgia (adults only): Grade 4 | 0 | 0 | 0 | 0
  Myalgia/Arthralgia (adults only): None reported/normal (temp) | 17 | 17 | 56 | 56
  Headache (adults only): Grade 1 | 3 | 4 | 0 | 0
  Headache (adults only): Grade 2 | 0 | 0 | 0 | 0
  Headache (adults only): Grade 3 | 0 | 0 | 0 | 0
  Headache (adults only): Grade 4 | 0 | 0 | 0 | 0
  Headache (adults only): None reported/normal (temp) | 14 | 13 | 56 | 56
  Decreased Appetite: Grade 1 | 0 | 0 | 7 | 6
  Decreased Appetite: Grade 2 | 0 | 0 | 0 | 0
  Decreased Appetite: Grade 3 | 0 | 0 | 0 | 0
  Decreased Appetite: Grade 4 | 0 | 0 | 0 | 0
  Decreased Appetite: None reported/normal (temp) | 17 | 17 | 49 | 50
  Pain (adults only): Grade 1 | 10 | 9 | 0 | 0
  Pain (adults only): Grade 2 | 0 | 0 | 0 | 0
  Pain (adults only): Grade 3 | 0 | 0 | 0 | 0
  Pain (adults only): Grade 4 | 0 | 0 | 0 | 0
  Pain (adults only): None reported/normal (temp) | 7 | 8 | 56 | 56
  Tenderness: Grade 1 | 6 | 8 | 10 | 11
  Tenderness: Grade 2 | 0 | 0 | 2 | 1
  Tenderness: Grade 3 | 0 | 0 | 0 | 0
  Tenderness: Grade 4 | 0 | 0 | 0 | 0
  Tenderness: None reported/normal (temp) | 11 | 9 | 44 | 44
  Redness: Grade 1 | 0 | 0 | 1 | 2
  Redness: Grade 2 | 0 | 0 | 0 | 0
  Redness: Grade 3 | 0 | 0 | 0 | 0
  Redness: Grade 4 | 0 | 0 | 0 | 0
  Redness: None reported/normal (temp) | 17 | 17 | 55 | 54
  Swelling: Grade 1 | 0 | 0 | 4 | 1
  Swelling: Grade 2 | 0 | 0 | 2 | 0
  Swelling: Grade 3 | 0 | 0 | 0 | 0
  Swelling: Grade 4 | 0 | 0 | 0 | 0
  Swelling: None reported/normal (temp) | 17 | 17 | 50 | 55
  Irritability (toddlers only): Grade 1 | 0 | 0 | 4 | 3
  Irritability (toddlers only): Grade 2 | 0 | 0 | 0 | 0
  Irritability (toddlers only): Grade 3 | 0 | 0 | 0 | 0
  Irritability (toddlers only): Grade 4 | 0 | 0 | 0 | 0
  Irritability (toddlers only): None reported/normal (temp) | 17 | 17 | 52 | 53

2. Primary Outcome: Infant Subjects Experiencing Local and Systemic Reactogenicity, by Severity: Vaccination 1
Description: Local and systemic reactogenicity of the study vaccine was evaluated for severity by toxicity grading scale (0 [none], 1 [mild], 2 [moderate], 3 [severe], 4 [potentially life threatening]) and relatedness to the vaccination. Injection site events were by definition considered related to study vaccine. Reactogenicity was monitored at the following times:
  * At 60 (± 15) minutes following primary vaccination
  * Daily by field workers during Days 1 to 6 post vaccination
  * In the clinic on 7 days (+3) following each vaccination (Visit 2, 4, and 6 for infants).
Time Frame: 7 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Infant--PCV 10: Injection of SIIL PCV 10 given on Day 0
- Infant--Prevenar 13: Injection of Prevenar 13 on Day 0
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 100 | 100
Participants
  Temperature: Grade 1 | 29 | 34
  Temperature: Grade 2 | 11 | 7
  Temperature: None | 60 | 59
  Irritability: Grade 1 | 33 | 29
  Irritability: Grade 2 | 4 | 2
  Irritability: None | 63 | 69
  Drowsiness: Grade 1 | 8 | 1
  Drowsiness: Grade 2 | 0 | 1
  Drowsiness: None | 92 | 98
  Decreased appetite: Grade 1 | 10 | 1
  Decreased appetite: Grade 2 | 0 | 1
  Decreased appetite: None | 90 | 98
  Tenderness at injection site: Grade 1 | 15 | 12
  Tenderness at injection site: Grade 2 | 4 | 5
  Tenderness at injection site: None | 81 | 83
  Erythema/redness at injection site: Grade 1 | 1 | 8
  Erythema/redness at injection site: Grade 2 | 0 | 1
  Erythema/redness at injection site: None | 99 | 91
  Induration/swelling at injection site: Grade 1 | 4 | 8
  Induration/swelling at injection site: Grade 2 | 0 | 2
  Induration/swelling at injection site: None | 96 | 90

3. Primary Outcome: Infant Subjects Experiencing Local and Systemic Reactogenicity, by Severity: Vaccination 2
Description: as for outcome 2
Time Frame: 7 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Infant--PCV 10: Injection of SIIL PCV 10 given on Days 0 and 28
- Infant--Prevenar 13: Injection of Prevenar 13 on Days 0 and 28
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 100 | 100
Participants
  Temperature: Grade 1 | 11 | 13
  Temperature: Grade 2 | 7 | 6
  Temperature: None | 82 | 81
  Irritability: Grade 1 | 35 | 30
  Irritability: Grade 2 | 5 | 3
  Irritability: None | 60 | 67
  Drowsiness: Grade 1 | 6 | 1
  Drowsiness: Grade 2 | 0 | 1
  Drowsiness: None | 94 | 98
  Decreased appetite: Grade 1 | 9 | 8
  Decreased appetite: Grade 2 | 1 | 0
  Decreased appetite: None | 90 | 92
  Tenderness at injection site: Grade 1 | 18 | 26
  Tenderness at injection site: Grade 2 | 2 | 1
  Tenderness at injection site: None | 80 | 73
  Erythema/redness at injection site: Grade 1 | 0 | 4
  Erythema/redness at injection site: Grade 2 | 1 | 1
  Erythema/redness at injection site: None | 99 | 95
  Induration/swelling at injection site: Grade 1 | 7 | 16
  Induration/swelling at injection site: Grade 2 | 1 | 2
  Induration/swelling at injection site: None | 92 | 82

4. Primary Outcome: Infant Subjects Experiencing Local and Systemic Reactogenicity, by Severity: Vaccination 3
Description: as for outcome 2
Time Frame: 7 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Infant--PCV 10: Injection of SIIL PCV 10 given on Days 0, 28, & 56.
- Infant--Prevenar 13: Injection of Prevenar 13 on Days 0, 28, & 56.
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 100 | 100
Participants
  Temperature: Grade 1 | 15 | 16
  Temperature: Grade 2 | 4 | 4
  Temperature: Grade 3 | 1 | 0
  Temperature: None | 80 | 80
  Irritability: Grade 1 | 33 | 37
  Irritability: Grade 2 | 3 | 4
  Irritability: Grade 3 | 1 | 0
  Irritability: None | 63 | 59
  Drowsiness: Grade 1 | 2 | 3
  Drowsiness: Grade 2 | 0 | 0
  Drowsiness: Grade 3 | 0 | 0
  Drowsiness: None | 98 | 97
  Decreased appetite: Grade 1 | 6 | 9
  Decreased appetite: Grade 2 | 1 | 2
  Decreased appetite: Grade 3 | 0 | 0
  Decreased appetite: None | 93 | 89
  Tenderness at injection site: Grade 1 | 21 | 19
  Tenderness at injection site: Grade 2 | 0 | 2
  Tenderness at injection site: Grade 3 | 0 | 0
  Tenderness at injection site: None | 79 | 79
  Erythema/redness at injection site: Grade 1 | 3 | 3
  Erythema/redness at injection site: Grade 2 | 0 | 0
  Erythema/redness at injection site: Grade 3 | 0 | 0
  Erythema/redness at injection site: None | 97 | 97
  Induration/swelling at injection site: Grade 1 | 11 | 13
  Induration/swelling at injection site: Grade 2 | 2 | 1
  Induration/swelling at injection site: Grade 3 | 0 | 0
  Induration/swelling at injection site: None | 87 | 86

5. Primary Outcome: Occurrence, Severity and Relatedness of All Adverse Events in Adults and Toddlers
Description: Reported here are only adverse events occurring in 5% or more of subjects; unless specifically stated, AEs were regarded as unrelated.
Time Frame: 28 days
Population: All subjects who received at least 1 study vaccination and had at least 1 post vaccination safety measurement and experienced an AE at a rate of 5% or more.
Measure: Count of Participants; unit: Participants
Groups:
- Adults--PCV 10; Toddler--PCV 10: Single dose of SIILPCV 10 at Day 0
- Adults--Pneumovax 23: Single dose of Pneumovax 23 at Day 0
- Toddler--Prevenar 13: Single dose of Prevenar 13 at Day 0
Arm/Group | Adults--PCV 10 | Adults--Pneumovax 23 | Toddler--PCV 10 | Toddler--Prevenar 13
Number analyzed (Participants) | 17 | 17 | 56 | 56
Participants
  Microcytic Anemia (Toddlers): Mild | 0 | 0 | 1 | 3
  Microcytic Anemia (Toddlers): Moderate | 0 | 0 | 0 | 1
  Microcytic Anemia (Toddlers): Severe | 0 | 0 | 2 | 0
  Microcytic Anemia (Toddlers): None | 17 | 17 | 53 | 52
  Diarrhea (Both): Mild | 0 | 1 | 7 | 5
  Diarrhea (Both): Moderate | 0 | 0 | 0 | 1
  Diarrhea (Both): Severe | 0 | 0 | 0 | 0
  Diarrhea (Both): None | 17 | 16 | 49 | 50
  Diarrhea--related: Mild | 0 | 0 | 1 | 0
  Diarrhea--related: Moderate | 0 | 0 | 0 | 0
  Diarrhea--related: Severe | 0 | 0 | 0 | 0
  Diarrhea--related: None | 17 | 17 | 55 | 56
  Pyrexia (Toddlers): Mild | 0 | 0 | 1 | 2
  Pyrexia (Toddlers): Moderate | 0 | 0 | 1 | 2
  Pyrexia (Toddlers): Severe | 0 | 0 | 0 | 0
  Pyrexia (Toddlers): None | 17 | 17 | 54 | 52
  Furuncle (Toddlers): Mild | 0 | 0 | 1 | 5
  Furuncle (Toddlers): Moderate | 0 | 0 | 0 | 0
  Furuncle (Toddlers): Severe | 0 | 0 | 0 | 0
  Furuncle (Toddlers): None | 17 | 17 | 55 | 51
  Gastroenteritis (Toddlers): Mild | 0 | 0 | 2 | 4
  Gastroenteritis (Toddlers): Moderate | 0 | 0 | 0 | 1
  Gastroenteritis (Toddlers): Severe | 0 | 0 | 1 | 0
  Gastroenteritis (Toddlers): None | 17 | 17 | 53 | 51
  Nasopharyngitis (Toddlers): Mild | 0 | 0 | 7 | 5
  Nasopharyngitis (Toddlers): Moderate | 0 | 0 | 0 | 0
  Nasopharyngitis (Toddlers): Severe | 0 | 0 | 0 | 0
  Nasopharyngitis (Toddlers): None | 17 | 17 | 49 | 51
  Tinea infection (Toddlers): Mild | 0 | 0 | 4 | 1
  Tinea infection (Toddlers): Moderate | 0 | 0 | 0 | 0
  Tinea infection (Toddlers): Severe | 0 | 0 | 0 | 0
  Tinea infection (Toddlers): None | 17 | 17 | 52 | 55
  Upper respiratory infection (Both): Mild | 1 | 1 | 6 | 7
  Upper respiratory infection (Both): Moderate | 0 | 0 | 2 | 2
  Upper respiratory infection (Both): Severe | 0 | 0 | 0 | 0
  Upper respiratory infection (Both): None | 16 | 16 | 48 | 47
  Abdominal pain (Adults): Mild | 1 | 3 | 0 | 0
  Abdominal pain (Adults): Moderate | 0 | 3 | 0 | 0
  Abdominal pain (Adults): Severe | 0 | 0 | 0 | 0
  Abdominal pain (Adults): None | 16 | 11 | 56 | 56
  Food poisoning (Adults): Mild | 0 | 0 | 0 | 0
  Food poisoning (Adults): Moderate | 0 | 1 | 0 | 0
  Food poisoning (Adults): Severe | 0 | 0 | 0 | 0
  Food poisoning (Adults): None | 17 | 16 | 56 | 56
  Toothache (Adults): Mild | 0 | 1 | 0 | 0
  Toothache (Adults): Moderate | 1 | 1 | 0 | 0
  Toothache (Adults): Severe | 0 | 0 | 0 | 0
  Toothache (Adults): None | 16 | 15 | 56 | 56
  Axillary pain (Adults): Mild | 1 | 1 | 0 | 0
  Axillary pain (Adults): Moderate | 0 | 0 | 0 | 0
  Axillary pain (Adults): Severe | 0 | 0 | 0 | 0
  Axillary pain (Adults): None | 16 | 16 | 56 | 56
  Axillary pain--related: Mild | 1 | 1 | 0 | 0
  Axillary pain--related: Moderate | 0 | 0 | 0 | 0
  Axillary pain--related: Severe | 0 | 0 | 0 | 0
  Axillary pain--related: None | 16 | 16 | 56 | 56
  Vaccination site pruritis (Both): Mild | 0 | 1 | 0 | 1
  Vaccination site pruritis (Both): Moderate | 0 | 0 | 0 | 0
  Vaccination site pruritis (Both): Severe | 0 | 0 | 0 | 0
  Vaccination site pruritis (Both): None | 17 | 16 | 56 | 55
  Vaccination site pruritis--related: Mild | 0 | 1 | 0 | 1
  Vaccination site pruritis--related: Moderate | 0 | 0 | 0 | 0
  Vaccination site pruritis--related: Severe | 0 | 0 | 0 | 0
  Vaccination site pruritis--related: None | 17 | 16 | 56 | 55
  Vaccination site swelling (Adults): Mild | 0 | 1 | 0 | 0
  Vaccination site swelling (Adults): Moderate | 0 | 0 | 0 | 0
  Vaccination site swelling (Adults): Severe | 0 | 0 | 0 | 0
  Vaccination site swelling (Adults): None | 17 | 16 | 56 | 56
  Vaccination site swelling--related: Mild | 0 | 1 | 0 | 0
  Vaccination site swelling--related: Moderate | 0 | 0 | 0 | 0
  Vaccination site swelling--related: Severe | 0 | 0 | 0 | 0
  Vaccination site swelling--related: None | 17 | 16 | 56 | 56
  Abscess (Adults): Mild | 0 | 0 | 0 | 0
  Abscess (Adults): Moderate | 0 | 1 | 0 | 0
  Abscess (Adults): Severe | 0 | 0 | 0 | 0
  Abscess (Adults): None | 17 | 16 | 56 | 56
  Otitis media (Adults): Mild | 1 | 0 | 0 | 0
  Otitis media (Adults): Moderate | 0 | 0 | 0 | 0
  Otitis media (Adults): Severe | 0 | 0 | 0 | 0
  Otitis media (Adults): None | 16 | 17 | 56 | 56
  Tonsillitis (Adults): Mild | 0 | 1 | 0 | 0
  Tonsillitis (Adults): Moderate | 0 | 0 | 0 | 0
  Tonsillitis (Adults): Severe | 0 | 0 | 0 | 0
  Tonsillitis (Adults): None | 17 | 16 | 56 | 56
  Urinary tract infection (Adults): Mild | 0 | 0 | 0 | 0
  Urinary tract infection (Adults): Moderate | 0 | 1 | 0 | 0
  Urinary tract infection (Adults): Severe | 0 | 0 | 0 | 0
  Urinary tract infection (Adults): None | 17 | 16 | 56 | 56
  Dizziness (Adults): Mild | 0 | 1 | 0 | 0
  Dizziness (Adults): Moderate | 1 | 0 | 0 | 0
  Dizziness (Adults): Severe | 0 | 0 | 0 | 0
  Dizziness (Adults): None | 16 | 16 | 56 | 56
  Dizziness--related: Mild | 0 | 1 | 0 | 0
  Dizziness--related: Moderate | 0 | 0 | 0 | 0
  Dizziness--related: Severe | 0 | 0 | 0 | 0
  Dizziness--related: None | 17 | 16 | 56 | 56

6. Primary Outcome: Occurrence, Severity and Relatedness of All Adverse Events in Infants
Description: Reported here are adverse events that occurred in 5% or more of the infant cohort. Booster dose safety results are reported separately. Unless stated, AEs are regarded as unrelated.
Time Frame: 12 weeks post last vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 100 | 100
Participants
  Diarrhea | 29 | 19
  Pyrexia | 9 | 3
  Vaccination site reaction (routine vaccines) | 11 | 4
  Vaccination site swelling (routine vaccines) | 55 | 61
  Vaccination site swelling (study vaccine) | 1 | 6
  Bronchiolitis | 5 | 6
  Conjunctivitis | 27 | 19
  Furuncle | 8 | 6
  Gastroenteritis | 13 | 10
  Impetigo | 5 | 4
  Nasopharyngitis | 19 | 17
  Otitis media--acute | 5 | 4
  Pneumonia | 8 | 8
  Tinea infection | 31 | 21
  Upper respiratory tract infection | 64 | 48
  Cough | 12 | 7
  Diaper dermatitis | 4 | 5
  Papular rash | 5 | 8
  Serious Adverse Event (SAE): Diarrhea | 1 | 0
  SAE: Gastroenteritis | 1 | 0
  SAE: Bronchiolitis | 3 | 1
  SAE: Atypical pneumonia | 1 | 0
  SAE: Sepsis | 0 | 1

7. Primary Outcome: Occurrence, Severity and Relatedness of Clinically Significant Hematological and Biochemistry Lab Values in Adults and Toddlers
Description: Blood samples were collected for safety hematology and clinical chemistry evaluations, organ function tests, and, for adults, coagulation panel evaluation. Laboratory assessments were only performed at baseline for infants. Testing for HIV was undertaken only following pre-test counseling of the subject/subject's parent as to the implications of the test result. Post test counseling was also undertaken, and on the basis of a positive result the subject and subject's parents would have been referred on for HIV care according to normal local practice in The Gambia.
Time Frame: 7 days after vaccination
Population: This table displays vaccinated adults and toddlers only. Infants had laboratory tests only at screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult SIILPCV10 | Adult Pneumovax 23 | Toddler SIILPCV10 | Toddler Prevenar 13
Number analyzed (Participants) | 17 | 17 | 56 | 56
Participants
  Decreased WBCs--not related: Mild | 0 | 0 | 0 | 0
  Decreased WBCs--not related: Moderate | 1 | 0 | 0 | 0
  Decreased WBCs--not related: Severe | 0 | 1 | 0 | 0
  Decreased WBCs--not related: None | 16 | 16 | 56 | 56
  Decreased WBCs--vaccine related: Mild | 0 | 0 | 0 | 0
  Decreased WBCs--vaccine related: Moderate | 0 | 1 | 0 | 0
  Decreased WBCs--vaccine related: Severe | 0 | 0 | 0 | 0
  Decreased WBCs--vaccine related: None | 17 | 16 | 56 | 56
  Increased WBCs--not related: Mild | 0 | 0 | 0 | 0
  Increased WBCs--not related: Moderate | 0 | 0 | 1 | 1
  Increased WBCs--not related: Severe | 0 | 0 | 0 | 0
  Increased WBCs--not related: None | 17 | 17 | 55 | 55
  Increased WBCs--vaccine related: Mild | 0 | 0 | 0 | 0
  Increased WBCs--vaccine related: Moderate | 0 | 0 | 1 | 0
  Increased WBCs--vaccine related: Severe | 0 | 0 | 0 | 0
  Increased WBCs--vaccine related: None | 17 | 17 | 55 | 56
  Decreased hemoglobin--not related: Mild | 0 | 0 | 0 | 0
  Decreased hemoglobin--not related: Moderate | 0 | 0 | 0 | 0
  Decreased hemoglobin--not related: Severe | 0 | 0 | 5 | 10
  Decreased hemoglobin--not related: None | 17 | 17 | 51 | 46
  Decreased hemoglobin--vaccine related: Mild | 0 | 0 | 0 | 0
  Decreased hemoglobin--vaccine related: Moderate | 0 | 0 | 0 | 0
  Decreased hemoglobin--vaccine related: Severe | 0 | 0 | 0 | 0
  Decreased hemoglobin--vaccine related: None | 17 | 17 | 56 | 56
  Increased ALT--not related: Mild | 0 | 0 | 0 | 0
  Increased ALT--not related: Moderate | 0 | 0 | 0 | 0
  Increased ALT--not related: Severe | 0 | 0 | 0 | 0
  Increased ALT--not related: None | 17 | 17 | 56 | 56
  Increased ALT--vaccine related: Mild | 0 | 0 | 1 | 0
  Increased ALT--vaccine related: Moderate | 0 | 0 | 0 | 0
  Increased ALT--vaccine related: Severe | 0 | 0 | 0 | 0
  Increased ALT--vaccine related: None | 17 | 17 | 55 | 56
  Decreased platelets--not related: Mild | 0 | 0 | 0 | 0
  Decreased platelets--not related: Moderate | 0 | 0 | 0 | 0
  Decreased platelets--not related: Severe | 0 | 0 | 0 | 0
  Decreased platelets--not related: None | 17 | 17 | 56 | 56
  Decreased platelets--vaccine related: Mild | 0 | 0 | 0 | 1
  Decreased platelets--vaccine related: Moderate | 0 | 0 | 0 | 0
  Decreased platelets--vaccine related: Severe | 0 | 0 | 0 | 0
  Decreased platelets--vaccine related: None | 17 | 17 | 56 | 55

8. Secondary Outcome: Geometric Mean Concentration of Immunoglobulin G (IgG) for Adults
Description: Serum samples were collected 28 days after the vaccination in adults to determine the ELISA IgG concentration for all 10 serotypes contained in SIILPCV10.
Time Frame: 4 weeks after vaccination
Population: All subjects who received the study vaccine per the assigned treatment group, and had post-dose immunogenicity measurement(s) with no major protocol violations that were determined to potentially interfere with immune response to the study vaccine.
Measure: Geometric Mean (90% Confidence Interval); unit: µg/mL
Arm/Group | Adults--PCV 10 | Adults--Pneumovax 23
Number analyzed (Participants) | 17 | 17
µg/mL
  PnC-IgG-ELISA type 1 | 3.96 [2.51 to 6.24] | 12.79 [8.34 to 19.61]
  PnC-IgG-ELISA type 5 | 3.56 [2.11 to 6.01] | 4.80 [3.07 to 7.51]
  PnC-IgG-ELISA type 6A: number analyzed (Participants) | 16 | 16
  PnC-IgG-ELISA type 6A | 17.09 [9.64 to 30.29] | 3.64 [2.59 to 5.12]
  PnC-IgG-ELISA type 6B: number analyzed (Participants) | 12 | 15
  PnC-IgG-ELISA type 6B | 26.87 [15.24 to 47.36] | 12.12 [8.12 to 18.07]
  PnC-IgG-ELISA type 7F | 4.62 [3.44 to 6.20] | 6.07 [4.10 to 9.0]
  PnC-IgG-ELISA type 9V | 4.92 [3.45 to 7.03] | 8.73 [6.70 to 11.37]
  PnC-IgG-ELISA type 14: number analyzed (Participants) | 14 | 16
  PnC-IgG-ELISA type 14 | 48.23 [31.60 to 73.62] | 44.78 [33.13 to 60.52]
  PnC-IgG-ELISA type 19A: number analyzed (Participants) | 17 | 16
  PnC-IgG-ELISA type 19A | 19.47 [12.13 to 31.25] | 11.20 [6.26 to 20.05]
  PnC-IgG-ELISA type 19F | 20.72 [14.62 to 29.37] | 12.38 [7.53 to 20.37]
  PnC-IgG-ELISA type 23F | 10.09 [6.26 to 16.24] | 8.95 [5.61 to 14.28]
Statistical Analysis 1: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — GMC will be summarized by treatment group with corresponding two-sided 90% CIs based on the t-distribution to provide population estimates; p = 0.0025, t-test, 2 sided; Pn IgG type 1 GMC Ratio = 0.31, 90% CI 2-sided [0.17 to 0.57]
Statistical Analysis 2: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.4540, t-test, 2 sided; Pn IgG type 5 GMC Ratio = 0.74, 90% CI 2-sided [0.38 to 1.45]
Statistical Analysis 3: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0003, t-test, 2 sided; Pn IgG type 6A GMC Ratio = 4.69, 90% CI 2-sided [2.46 to 8.94]
Statistical Analysis 4: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0460, t-test, 2 sided; Pn IgG type 6B GMC Ratio = 2.22, 90% CI 2-sided [1.16 to 4.24]
Statistical Analysis 5: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.3365, t-test, 2 sided; Pn IgG type 7F GMC Ratio = 0.76, 90% CI 2-sided [0.47 to 1.22]
Statistical Analysis 6: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0313, t-test, 2 sided; Pn IgG type 9V GMC Ratio = 0.56, 90% CI 2-sided [0.37 to 0.87]
Statistical Analysis 7: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.8060, t-test, 2 sided; Pn IgG type 14 GMC Ratio = 1.08, 90% CI 2-sided [0.65 to 1.79]
Statistical Analysis 8: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.2044, t-test, 2 sided; Pn IgG type 19A GMC Ratio = 1.74, 90% CI 2-sided [0.84 to 3.58]
Statistical Analysis 9: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.1490, t-test, 2 sided; Pn IgG type 19F GMC Ratio = 1.67, 90% CI 2-sided [0.93 to 3.02]
Statistical Analysis 10: Comparison: Adults--PCV 10 vs Adults--Pneumovax 23; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.7565, t-test, 2 sided; Pn IgG type 23F GMC Ratio = 1.13, 90% CI 2-sided [0.59 to 2.15]

9. Secondary Outcome: Geometric Mean Concentration of Immunoglobulin G (IgG) 4 Weeks After Vaccination for Toddlers
Description: Serum samples were collected 28 days after vaccination for toddlers to determine the ELISA IgG concentration for all 10 serotypes contained in SIILPCV10.
Time Frame: 4 weeks after vaccination
Population: as for outcome 8
Measure: Geometric Mean (90% Confidence Interval); unit: µg/mL
Groups:
- Toddler--PCV 10: Dose of SIILPCV 10 on Day 0
- Toddler--Prevenar 13: Dose of Prevenar 13 on Day 0
Arm/Group | Toddler--PCV 10 | Toddler--Prevenar 13
Number analyzed (Participants) | 56 | 56
µg/mL
  PnC-IgG-ELISA type 1: Baseline | 0.77 [0.46 to 1.36] | 0.92 [0.72 to 1.26]
  PnC-IgG-ELISA type 1: Post-vaccination | 4.59 [4.03 to 5.67] | 6.09 [4.93 to 10.17]
  PnC-IgG-ELISA type 5: Baseline | 0.60 [0.36 to 1.04] | 0.42 [0.32 to 0.51]
  PnC-IgG-ELISA type 5: Post-vaccination | 2.30 [1.67 to 3.48] | 3.35 [2.63 to 5.03]
  PnC-IgG-ELISA type 6A: Baseline | 1.40 [0.88 to 2.67] | 1.29 [0.97 to 1.72]
  PnC-IgG-ELISA type 6A: Post-vaccination | 13.33 [10.15 to 20.81] | 15.83 [12.52 to 25.12]
  PnC-IgG-ELISA type 6B: Baseline | 2.02 [1.29 to 3.42] | 1.95 [1.41 to 2.55]
  PnC-IgG-ELISA type 6B: Post-vaccination | 15.77 [12.20 to 22.43] | 19.16 [15.81 to 28.72]
  PnC-IgG-ELISA type 7F: Baseline | 1.49 [0.96 to 2.10] | 1.46 [0.99 to 1.86]
  PnC-IgG-ELISA type 7F: Post-vaccination | 9.17 [7.69 to 11.64] | 12.35 [9.41 to 18.55]
  PnC-IgG-ELISA type 9V: Baseline | 0.53 [0.31 to 0.86] | 0.41 [0.28 to 0.51]
  PnC-IgG-ELISA type 9V: Post-vaccination | 2.35 [1.69 to 3.25] | 3.90 [2.79 to 5.95]
  PnC-IgG-ELISA type 14: Baseline | 2.89 [1.60 to 4.40] | 2.47 [1.70 to 3.80]
  PnC-IgG-ELISA type 14: Post-vaccination | 14.55 [9.29 to 20.60] | 8.28 [6.49 to 12.55]
  PnC-IgG-ELISA type 19A: Baseline | 1.17 [0.63 to 1.97] | 0.57 [0.34 to 0.72]
  PnC-IgG-ELISA type 19A: Post-vaccination | 9.76 [7.23 to 12.18] | 13.68 [7.12 to 20.02]
  PnC-IgG-ELISA type 19F: Baseline | 1.75 [0.85 to 3.43] | 0.97 [0.65 to 1.58]
  PnC-IgG-ELISA type 19F: Post-vaccination | 9.75 [7.76 to 12.26] | 12.87 [9.08 to 20.75]
  PnC-IgG-ELISA type 23F: Baseline | 0.71 [0.39 to 1.32] | 0.63 [0.44 to 1.05]
  PnC-IgG-ELISA type 23F: Post-vaccination | 6.84 [4.76 to 10.03] | 10.49 [8.21 to 18.16]
Statistical Analysis 1: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — GMC will be summarized by treatment group with corresponding two-sided 90% CIs based on the t-distribution to provide population estimates. Due to distributional characteristics, confidence intervals around GMCs and treatment-group ratio are estimated using bootstrap resampling (10,000 bootstrap samples); p = 0.2653, Two-tailed from z-test; Pn IgG type 1 GMC Ratio = 0.75, 90% CI 2-sided [0.54 to 1.31]
Statistical Analysis 2: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.2059, Two-tailed from z-test; Pn IgG type 5 GMC Ratio = 0.69, 90% CI 2-sided [0.45 to 1.20]
Statistical Analysis 3: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.5664, Two-tailed from z-test; Pn IgG type 6A GMC Ratio = 0.84, 90% CI 2-sided [0.55 to 1.54]
Statistical Analysis 4: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.4456, Two-tailed from z-test; Pn IgG type 6B GMC Ratio = 0.82, 90% CI 2-sided [0.57 to 1.31]
Statistical Analysis 5: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.2189, Two-tailed from z-test; Pn IgG type 7F GMC Ratio = 0.74, 90% CI 2-sided [0.52 to 1.14]
Statistical Analysis 6: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0970, Two-tailed from z-test; Pn IgG type 9V GMC Ratio = 0.60, 90% CI 2-sided [0.38 to 1.03]
Statistical Analysis 7: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0713, Two-tailed from z-test; Pn IgG type 14 GMC Ratio = 1.76, 90% CI 2-sided [1.02 to 2.79]
Statistical Analysis 8: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.3443, Two-tailed from z-test; Pn IgG type 19A GMC Ratio = 0.71, 90% CI 2-sided [0.42 to 1.35]
Statistical Analysis 9: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.3278, Two-tailed from z-test; Pn IgG type 19F GMC Ratio = 0.76, 90% CI 2-sided [0.48 to 1.23]
Statistical Analysis 10: Comparison: Toddler--PCV 10 vs Toddler--Prevenar 13; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.2039, Two-tailed from z-test; Pn IgG type 23F GMC Ratio = 0.65, 90% CI 2-sided [0.40 to 1.16]

10. Secondary Outcome: Geometric Mean Concentration of Immunoglobulin G (IgG) 4 Weeks After Vaccination for Infants
Description: Serum samples were collected 28 days after the third vaccination for infants to determine the ELISA IgG concentration for all 10 serotypes contained in SIILPCV10.
Time Frame: 4 weeks after the third dose
Population: All subjects who received all study vaccines per the assigned treatment group, and had post-dose immunogenicity measurement(s) with no major protocol violations that were determined to potentially interfere with immune response to the study vaccine.
Measure: Geometric Mean (90% Confidence Interval); unit: µg/mL
Groups:
- Infant--PCV 10: Dose of SIILPCV 10 on Day 0, 28 and 56
- Infant--Prevenar 13: Dose of Prevenar 13 on Day 0, 28 and 56
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 100 | 100
µg/mL
  PnC-IgG-ELISA type 1 | 2.99 [2.61 to 3.43] | 3.38 [3.02 to 3.78]
  PnC-IgG-ELISA type 5 | 2.09 [1.86 to 2.36] | 1.74 [1.53 to 1.98]
  PnC-IgG-ELISA type 6A | 1.02 [0.83 to 1.27] | 1.82 [1.53 to 2.17]
  PnC-IgG-ELISA type 6B: number analyzed (Participants) | 100 | 96
  PnC-IgG-ELISA type 6B | 1.57 [1.28 to 1.92] | 3.64 [3.01 to 4.42]
  PnC-IgG-ELISA type 7F | 2.19 [1.89 to 2.53] | 3.88 [3.44 to 4.38]
  PnC-IgG-ELISA type 9V | 1.07 [0.93 to 1.23] | 2.19 [1.91 to 2.50]
  PnC-IgG-ELISA type 14: number analyzed (Participants) | 100 | 99
  PnC-IgG-ELISA type 14 | 4.96 [4.20 to 5.87] | 4.47 [3.62 to 5.53]
  PnC-IgG-ELISA type 19A: number analyzed (Participants) | 100 | 96
  PnC-IgG-ELISA type 19A | 1.49 [1.26 to 1.76] | 5.20 [4.37 to 6.20]
  PnC-IgG-ELISA type 19F: number analyzed (Participants) | 100 | 96
  PnC-IgG-ELISA type 19F | 3.87 [3.35 to 4.49] | 5.38 [4.79 to 6.05]
  PnC-IgG-ELISA type 23F | 1.56 [1.32 to 1.83] | 2.68 [2.28 to 3.15]
Statistical Analysis 1: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.2550, t-test, 2 sided; Pn IgG type 1 GMC Ratio = 0.89, 90% CI 2-sided [0.74 to 1.06]
Statistical Analysis 2: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0865, t-test, 2 sided; Pn IgG type 5 GMC Ratio = 1.20, 90% CI 2-sided [1.01 to 1.43]
Statistical Analysis 3: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0006, t-test, 2 sided; Pn IgG type 6A GMC Ratio = 0.56, 90% CI 2-sided [0.43 to 0.74]
Statistical Analysis 4: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.0001, t-test, 2 sided; Pn IgG type 6B GMC Ratio = 0.43, 90% CI 2-sided [0.33 to 0.57]
Statistical Analysis 5: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.0001, t-test, 2 sided; Pn IgG type 7F GMC Ratio = 0.56, 90% CI 2-sided [0.47 to 0.68]
Statistical Analysis 6: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.0001, t-test, 2 sided; Pn IgG type 9V GMC Ratio = 0.49, 90% CI 2-sided [0.41 to 0.59]
Statistical Analysis 7: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.5234, t-test, 2 sided; Pn IgG type 14 GMC Ratio = 1.11, 90% CI 2-sided [0.85 to 1.45]
Statistical Analysis 8: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p < 0.0001, t-test, 2 sided; Pn IgG type 19A GMC Ratio = 0.29, 90% CI 2-sided [0.22 to 0.36]
Statistical Analysis 9: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0040, t-test, 2 sided; Pn IgG type 19F GMC Ratio = 0.72, 90% CI 2-sided [0.60 to 0.87]
Statistical Analysis 10: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0001, t-test, 2 sided; Pn IgG type 23F GMC Ratio = 0.58, 90% CI 2-sided [0.46 to 0.73]

11. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Immunoglobulin G (IgG) in Toddlers, by Serotype
Description: Serum samples were collected before the first vaccination and 28 days after the last vaccination for adults and toddlers and 28 days after the completion of the primary series for infants to determine the ELISA IgG concentration for all 10 serotypes contained in SIILPCV10. Blood samples were also collected for immunogenicity testing before and 28 days after the booster dose for infants. Baseline serum samples for infants and adults were not assayed. The IgG concentration was also determined for each component of the co administered pentavalent vaccine (DTwP-HepB-Hib) in sera from the infant cohort. If there were limitations to blood volumes, appropriate subsets and priorities for immune testing were established with the immunology laboratories to ensure measurements were unbiased and representative of the entire cohort.
Time Frame: 4 weeks after vaccination (28 days)
Population: The evaluable group differs for individual serotypes due to non-reportable results.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Arm/Group | Toddler--PCV 10 | Toddler--Prevenar 13
Number analyzed (Participants) | 17 | 17
fold change
  PnC-IgG-ELISA type 1 | 5.99 [3.94 to 10.12] | 6.59 [5.06 to 11.10]
  PnC-IgG-ELISA type 5 | 3.82 [2.67 to 6.67] | 8.00 [6.79 to 12.16]
  PnC-IgG-ELISA type 6A | 9.91 [6.14 to 19.88] | 12.31 [9.81 to 20.31]
  PnC-IgG-ELISA type 6B | 7.79 [5.02 to 14.78] | 9.82 [8.12 to 15.03]
  PnC-IgG-ELISA type 7F | 6.16 [4.68 to 9.94] | 8.44 [6.83 to 13.90]
  PnC-IgG-ELISA type 9V | 4.43 [3.30 to 6.93] | 9.58 [7.81 to 15.35]
  PnC-IgG-ELISA type 14 | 5.04 [3.52 to 7.42] | 3.35 [2.41 to 5.12]
  PnC-IgG-ELISA type 19A | 7.89 [4.56 to 15.32] | 24.17 [18.51 to 36.37]
  PnC-IgG-ELISA type 19F | 5.73 [3.24 to 13.28] | 13.26 [9.35 to 21.82]
  PnC-IgG-ELISA type 23F | 9.67 [6.11 to 17.18] | 16.54 [12.53 to 28.13]

12. Secondary Outcome: Number and Percentage of Immunoglobulin G (IgG) Seroresponders Among Infants, by Serotype
Description: Seroresponse was defined as ≥ 0.35 µg/mL. In infants, serum samples were collected 28 days after receipt of three doses of the vaccine to determine the ELISA IgG concentration for all 10 serotypes contained in SIILPCV10.
Time Frame: 4 weeks after third dose
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- Infant--PCV 10: Dose of SIILPCV 10 on Days 0, 28 & 56
- Infant--Prevenar 13: Dose of Prevenar 13 on Days 0, 28, & 56
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 100 | 100
Participants
  Pn-IgG-ELISA type 1 | 99 | 100
  Pn-IgG-ELISA type 5 | 100 | 97
  Pn-IgG-ELISA type 6A | 79 | 91
  Pn-IgG-ELISA type 6B | 89 | 93
  Pn-IgG-ELISA type 7F | 97 | 100
  Pn-IgG-ELISA type 9V | 94 | 97
  Pn-IgG-ELISA type 14 | 98 | 96
  Pn-IgG-ELISA type 19A | 92 | 94
  Pn-IgG-ELISA type 19F | 99 | 97
  Pn-IgG-ELISA type 23F | 91 | 97
Statistical Analysis 1: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — Treatment group differences were estimated by the difference in proportion of seroresponders, with 2-sided exact 90% CIs around the difference calculated using the unconditional exact method of Newcombe. Although inference regarding seroresponse was not of primary concern in this study, a 2-sided 90% CI that excluded 0 was indicative of statistically significant difference at p ≤ 0.10 not corrected for multiplicity analysis; Absolute Difference for Type 1 = -1.0, 90% CI 2-sided [-5.13 to 2.66]
Statistical Analysis 2: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 5 = 3.0, 90% CI 2-sided [-1.10 to 7.95]
Statistical Analysis 3: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 6A = -12.0, 90% CI 2-sided [-20.94 to -2.97]
Statistical Analysis 4: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 6B = -7.9, 90% CI 2-sided [-15.0 to -1.01]
Statistical Analysis 5: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 7F = -3.0, 90% CI 2-sided [-7.95 to 1.10]
Statistical Analysis 6: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 9V = -3.0, 90% CI 2-sided [-9.17 to 2.90]
Statistical Analysis 7: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 14 = 1.00, 90% CI 2-sided [-4.00 to 6.27]
Statistical Analysis 8: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 19A = -5.9, 90% CI 2-sided [-12.38 to 0.17]
Statistical Analysis 9: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 19F = 0.0, 90% CI 2-sided [-4.22 to 4.33]
Statistical Analysis 10: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 12, analysis 1]; Absolute Difference for Type 23F = -6.0, 90% CI 2-sided [-12.77 to 0.40]

13. Secondary Outcome: Functional Antibody (OPA) Geometric Mean Titers
Description: The functional activity of the IgG response to the 10 serotypes contained in SIILPCV10 was determined in randomly selected subsets of the infant and toddler cohorts and all adult subjects in the same serum samples collected 28 days after the last vaccinations. This activity was determined using the 4-fold multiplexed OPA developed at the University of Alabama at Birmingham.
Time Frame: 4 weeks after last vaccination
Population: Randomly selected subsets of the infant and toddler cohorts and all adult subjects
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Adults--PCV 10 | Adults--Pneumovax 23 | Toddler--PCV 10 | Toddler--Prevenar 13 | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 20 | 20
titer
  MOPA - Pn 1 | 18.89 [10.14 to 45.59] | 85.89 [43.15 to 215.84] | 436.31 [365.08 to 582.46] | 438.14 [278.73 to 890.17] | 50.65 [27.91 to 96.55] | 29.42 [15.58 to 68.08]
  MOPA - Pn 5 | 263.06 [138.91 to 499.28] | 265.56 [143.22 to 521.05] | 1358.22 [960.34 to 2087.48] | 1148.43 [929.92 to 1708.67] | 113.92 [74.12 to 167.10] | 104.83 [64.11 to 181.22]
  MOPA - Pn 6A | 17161.52 [12378.36 to 23946.20] | 4925.68 [3204.91 to 7661.38] | 19371.45 [12538.18 to 34268.51] | 12001.09 [8229.26 to 21545.31] | 1243.88 [942.40 to 1834.30] | 3068.16 [2267.85 to 5318.41]
  MOPA - 6B | 13303.68 [9432.51 to 18190.05] | 4221.68 [2890.62 to 5925.09] | 8768.08 [5471.57 to 12932.67] | 7066.76 [4456.49 to 11894.25] | 1530.37 [935.24 to 2368.41] | 2267.44 [1175.92 to 3718.87]
  MOPA - 7F | 7099.73 [4147.20 to 11222.44] | 8019.15 [4956.82 to 10917.82] | 10723.98 [7151.48 to 16590.09] | 12737.21 [8063.57 to 18328.98] | 876.58 [616.90 to 1221.31] | 3763.17 [2754.89 to 5393.72]
  MOPA - 9V | 3928.12 [2827.41 to 5629.89] | 4443.95 [3275.91 to 6299.32] | 3770.19 [2004.45 to 6384.49] | 4862.30 [3128.56 to 6953.05] | 197.24 [95.09 to 347.56] | 752.77 [528.18 to 1024.26]
  MOPA - 14 | 9148.12 [6271.81 to 12407.65] | 6707.26 [5098.03 to 7886.64] | 8213.23 [4526.63 to 13664.12] | 2557.27 [1597.17 to 3868.34] | 1243.39 [743.97 to 1912.05] | 1108.02 [501.79 to 2097.51]
  MOPA - 19A | 3170.33 [1906.55 to 4427.88] | 2215.22 [1314.65 to 3458.76] | 1789.98 [651.04 to 3498.32] | 3780.56 [2358.04 to 6045.56] | 151.31 [64.25 to 233.45] | 765.71 [589.49 to 886.28]
  MOPA - 19F | 3564.32 [2636.19 to 4898.79] | 2481.47 [1623.91 to 3860.16] | 3036.60 [2134.81 to 5126.44] | 3371.52 [2238.81 to 5853.53] | 744.92 [607.87 to 941.74] | 498.98 [275.77 to 723.41]
  MOPA - 23F | 5035.73 [3417.87 to 7587.87] | 2844.04 [2123.33 to 3737.09] | 12415.92 [8018.97 to 19342.91] | 10517.81 [5848.87 to 19460.60] | 627.27 [341.95 to 975.77] | 921.43 [574.79 to 1419.94]

14. Secondary Outcome: Number and Percentage of Functional (OPA) Infant Seroresponders, by Serotype
Description: The functional activity of the immune response to the 10 serotypes contained in SIILPCV10 was determined in randomly selected subsets of the infant cohort in the same serum samples collected 28 days after the completion of the primary series. This activity was determined using the 4-fold multiplexed OPA developed at the University of Alabama at Birmingham.
Time Frame: 84 days
Population: Randomly selected subsets of the infant cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 20 | 20
Participants
  MOPA - Pn 1: number analyzed (Participants) | 16 | 13
  MOPA - Pn 1 | 15 | 11
  MOPA - Pn 5 | 19 | 19
  MOPA - Pn 6A: number analyzed (Participants) | 20 | 19
  MOPA - Pn 6A | 20 | 18
  MOPA - 6B: number analyzed (Participants) | 19 | 20
  MOPA - 6B | 19 | 19
  MOPA - 7F | 20 | 20
  MOPA - 9V | 20 | 20
  MOPA - 14: number analyzed (Participants) | 19 | 19
  MOPA - 14 | 19 | 18
  MOPA - 19A: number analyzed (Participants) | 17 | 20
  MOPA - 19A | 16 | 20
  MOPA - 19F | 20 | 19
  MOPA - 23F | 20 | 20
Statistical Analysis 1: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — Exact confidence intervals around treatment group differences are calculated based on Newcombe score. Calculation of difference and confidence interval around the difference is not possible when all subjects in both groups are responders; Absolute difference for MOPA type 1 = 9.1, 90% CI 2-sided [-15.55 to 36.11]
Statistical Analysis 2: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 14, analysis 1]; Absolute difference for MOPA type 5 = 0.0, 90% CI 2-sided [-18.56 to 18.56]
Statistical Analysis 3: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 14, analysis 1]; Absolute difference for MOPA type 6B = 5.0, 90% CI 2-sided [-12.35 to 22.97]
Statistical Analysis 4: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 14, analysis 1]; Absolute difference for MOPA type 14 = 5.3, 90% CI 2-sided [-12.15 to 24.01]
Statistical Analysis 5: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 14, analysis 1]; Absolute difference for MOPA type 19A = -5.9, 90% CI 2-sided [-26.41 to 11.01]
Statistical Analysis 6: Comparison: Infant--PCV 10 vs Infant--Prevenar 13; Test type: Other — [test comment as in outcome 14, analysis 1]; Absolute difference for MOPA type 19F = 5.0, 90% CI 2-sided [-11.64 to 22.97]

15. Secondary Outcome: Number and Percentage of Immunoglobulin G (IgG) Seroresponders Against Pentavalent Vaccine Components
Description: Serum samples were collected 28 days after the third vaccination for infants to determine the ELISA IgG concentration for each component of the co administered pentavalent vaccine (DTwP-HepB-Hib) . Seroresponse was defined as equal to or greater concentrations for:
  * Diptheria toxoid: 0.1 IU/mL
  * Hepatitis B: 10 milli-International unit (mIU) /mL
  * Hib: 0.15 mcg/mL
  * Tetanus toxoid: 0.1 IU/mL
Time Frame: 84 days
Population: All subjects who receive all study vaccines per the assigned treatment group, and had post-dose immunogenicity measurement(s) with no major protocol violations that were determined to potentially interfere with immune response to the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 100 | 100
Participants
  Diphtheria toxoid | 100 | 100
  Hepatitis B | 100 | 100
  Hib (anti-PRP antibodies) | 100 | 99
  Tetanus toxoid | 100 | 100

16. Other Pre Specified Outcome: Infant Subjects Experiencing Local and Systemic Reactogenicity After Booster Vaccination, by Severity
Description: Local and systemic reactogenicity of the study vaccine was evaluated for severity by toxicity grading scale (0 [none], 1 [mild], 2 [moderate], 3 [severe], 4 [potentially life threatening]) and relatedness to the vaccination. Injection site events were by definition considered related to study vaccine. Reactogenicity was monitored at the following times:
  * At 30 (± 10) minutes following booster vaccination
  * Daily by field workers during Days 1 to 6 post vaccination
  * In the clinic on 7 days (+3) following the vaccination
Time Frame: 7 days
Population: A subset of the infant cohort who were eligible for the booster phase, had not yet received the Prevenar 13 booster that was offered to infants in the SIILPCV10 group as part of the primary phase of the study and who contributed at least some safety and/or immunogenicity data.
Measure: Count of Participants; unit: Participants
Groups:
- Infant--PCV 10: Booster injection of SIILPCV 10 at 9 months of age
- Prevenar 13: Booster injection of Prevenar 13 at 9 months of age
Arm/Group | Infant--PCV 10 | Prevenar 13
Number analyzed (Participants) | 49 | 47
Participants
  Temperature above 37 C: Grade 1 | 3 | 4
  Temperature above 37 C: Grade 2 | 1 | 1
  Temperature above 37 C: Grade 3 | 2 | 1
  Temperature above 37 C: Grade 4 | 0 | 0
  Temperature above 37 C: None reported/normal (temp) | 43 | 41
  Cutaneous Rash: Grade 1 | 1 | 3
  Cutaneous Rash: Grade 2 | 0 | 2
  Cutaneous Rash: Grade 3 | 0 | 0
  Cutaneous Rash: Grade 4 | 0 | 0
  Cutaneous Rash: None reported/normal (temp) | 48 | 42
  Irritability: Grade 1 | 5 | 7
  Irritability: Grade 2 | 0 | 0
  Irritability: Grade 3 | 0 | 0
  Irritability: Grade 4 | 0 | 0
  Irritability: None reported/normal (temp) | 44 | 40
  Drowsiness: Grade 1 | 0 | 1
  Drowsiness: Grade 2 | 1 | 0
  Drowsiness: Grade 3 | 0 | 0
  Drowsiness: Grade 4 | 0 | 0
  Drowsiness: None reported/normal (temp) | 48 | 46
  Decreased appetite: Grade 1 | 2 | 5
  Decreased appetite: Grade 2 | 0 | 0
  Decreased appetite: Grade 3 | 0 | 0
  Decreased appetite: Grade 4 | 0 | 0
  Decreased appetite: None reported/normal (temp) | 47 | 42
  Injection site tenderness: Grade 1 | 8 | 11
  Injection site tenderness: Grade 2 | 1 | 0
  Injection site tenderness: Grade 3 | 0 | 0
  Injection site tenderness: Grade 4 | 0 | 0
  Injection site tenderness: None reported/normal (temp) | 40 | 36
  Erythema: Grade 1 | 1 | 1
  Erythema: Grade 2 | 0 | 0
  Erythema: Grade 3 | 0 | 0
  Erythema: Grade 4 | 0 | 0
  Erythema: None reported/normal (temp) | 48 | 46
  Induration/Swelling: Grade 1 | 4 | 4
  Induration/Swelling: Grade 2 | 2 | 0
  Induration/Swelling: Grade 3 | 0 | 0
  Induration/Swelling: Grade 4 | 0 | 0
  Induration/Swelling: None reported/normal (temp) | 43 | 43

17. Other Pre Specified Outcome: Occurrence of All Adverse Events (AEs) and SAEs Following a Booster Vaccination Among Infants, by Type and Severity
Description: Unsolicited adverse events following a booster dose of SIILPCV10 occurring in 5% or greater of study participants. Unless specifically stated, AEs are considered unrelated.
Time Frame: 4 weeks (28 days)
Population: A subset of the infant cohort PP_IMM who were eligible for the booster phase, had not yet received the Prevenar 13 booster that was offered to infants in the SIILPCV10 group as part of the primary phase of the study and who contributed at least some safety and/or immunogenicity data.
Measure: Count of Participants; unit: Participants
Groups:
- Infant--PCV 10: Booster dose of SIILPCV 10 at 10 months of age
- Prevenar 13: Booster dose of Prevenar 13 at 10 months of age
Arm/Group | Infant--PCV 10 | Prevenar 13
Number analyzed (Participants) | 49 | 47
Participants
  Upper respiratory tract infection: Grade 1 | 14 | 6
  Upper respiratory tract infection: Grade 2 | 0 | 0
  Upper respiratory tract infection: Grade 3 | 0 | 0
  Upper respiratory tract infection: Grade 4 | 0 | 0
  Upper respiratory tract infection: None reported | 35 | 41
  Dermatitis: Grade 1 | 4 | 3
  Dermatitis: Grade 2 | 0 | 0
  Dermatitis: Grade 3 | 0 | 0
  Dermatitis: Grade 4 | 0 | 0
  Dermatitis: None reported | 45 | 44
  Diarrhea: Grade 1 | 2 | 5
  Diarrhea: Grade 2 | 0 | 0
  Diarrhea: Grade 3 | 0 | 0
  Diarrhea: Grade 4 | 0 | 0
  Diarrhea: None reported | 47 | 42
  Impetigo: Grade 1 | 3 | 3
  Impetigo: Grade 2 | 0 | 0
  Impetigo: Grade 3 | 0 | 0
  Impetigo: Grade 4 | 0 | 0
  Impetigo: None reported | 46 | 44
  Rash pustular: Grade 1 | 1 | 4
  Rash pustular: Grade 2 | 0 | 0
  Rash pustular: Grade 3 | 0 | 0
  Rash pustular: Grade 4 | 0 | 0
  Rash pustular: None reported | 48 | 43
  Pyrexia: Grade 1 | 1 | 3
  Pyrexia: Grade 2 | 0 | 0
  Pyrexia: Grade 3 | 0 | 0
  Pyrexia: Grade 4 | 0 | 0
  Pyrexia: None reported | 48 | 44
  SAE--severe malaria with severe anemia: Grade 1 | 0 | 0
  SAE--severe malaria with severe anemia: Grade 2 | 0 | 0
  SAE--severe malaria with severe anemia: Grade 3 | 1 | 0
  SAE--severe malaria with severe anemia: Grade 4 | 0 | 0
  SAE--severe malaria with severe anemia: None reported | 48 | 47

18. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) of Immunoglobulin G (IgG) by Time Point (4 Weeks Post Vaccination 3, Pre Booster, 4 Weeks Post Booster) Among Infants Receiving Booster Dose
Description: Using enzyme-linked immunosorbent assay (ELISA). Blood samples were collected for immunogenicity testing at 4 weeks post vaccination 3, and before and 28 days after the booster dose for infants.
Time Frame: 4 weeks (28 days)
Population: This is the population of infants who received a booster dose of either PCV-10 or Prevenar-13. The evaluable group differs for individual serotypes due to NR results.
Measure: Geometric Mean (90% Confidence Interval); unit: µg/mL
Groups:
- Infant--Prevenar 13: Booster dose of Prevenar 13 at 10 months of age
- Treatment Comparison (GMC Ratio): This column is the GMC Ratio between the SIILPCV 10 and the Prevenar 13 groups
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13 | Treatment Comparison (GMC Ratio)
Number analyzed (Participants) | 49 | 47 | 96
µg/mL
  PnC-IgG-ELISA Type 1: 4 weeks post Vac 3 | 2.67 [2.22 to 3.21] | 3.23 [2.76 to 3.78] | 0.83 [0.65 to 1.05]
  PnC-IgG-ELISA Type 1: Pre Booster | 0.27 [0.22 to 0.33] | 0.32 [0.27 to 0.40] | 0.83 [0.63 to 1.10]
  PnC-IgG-ELISA Type 1: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 1: Post Booster | 6.24 [4.62 to 8.42] | 5.11 [3.96 to 6.60] | 1.22 [0.83 to 1.81]
  PnC-IgG-ELISA Type 5: 4 weeks post Vac 3 | 2.01 [1.70 to 2.38] | 1.45 [1.18 to 1.79] | 1.38 [1.06 to 1.80]
  PnC-IgG-ELISA Type 5: Pre Booster | 0.16 [0.13 to 0.18] | 0.25 [0.21 to 0.30] | 0.62 [0.48 to 0.78]
  ELISA Type 5: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  ELISA Type 5: Post Booster | 2.30 [1.88 to 2.81] | 2.57 [2.10 to 3.13] | 0.90 [0.68 to 1.19]
  PnC-IgG-ELISA Type 6A: 4 weeks post Vac 3 | 1.06 [0.80 to 1.42] | 1.56 [1.17 to 2.06] | 0.68 [0.46 to 1.02]
  PnC-IgG-ELISA Type 6A: Pre Booster | 0.46 [0.38 to 0.56] | 0.53 [0.43 to 0.66] | 0.87 [0.65 to 1.16]
  PnC-IgG-ELISA Type 6A: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 6A: Post Booster | 9.50 [6.94 to 12.99] | 12.06 [9.98 to 14.56] | 0.79 [0.55 to 1.13]
  PnC-IgG-ELISA Type 6B: 4 weeks post Vac 3 | 1.39 [1.03 to 1.87] | 3.67 [2.74 to 4.93] | 0.38 [0.25 to 0.57]
  PnC-IgG-ELISA Type 6B: Pre Booster | 0.73 [0.59 to 0.90] | 0.50 [0.42 to 0.60] | 1.45 [1.10 to 1.90]
  PnC-IgG-ELISA Type 6B: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 6B: Post Booster | 12.72 [9.79 to 16.54] | 14.06 [11.55 to 17.11] | 0.91 [0.65 to 1.26]
  PnC-IgG-ELISA Type 7F: 4 weeks post Vac 3 | 1.99 [1.59 to 2.49] | 3.43 [2.81 to 4.18] | 0.58 [0.43 to 0.78]
  PnC-IgG-ELISA Type 7F: Pre Booster | 0.49 [0.39 to 0.62] | 0.81 [0.68 to 0.97] | 0.61 [0.45 to 0.81]
  PnC-IgG-ELISA Type 7F: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 7F: Post Booster | 6.76 [5.49 to 8.32] | 8.51 [7.05 to 10.26] | 0.79 [0.60 to 1.05]
  PnC-IgG-ELISA Type 9V: 4 weeks post Vac 3 | 1.06 [0.89 to 1.26] | 2.22 [1.84 to 2.68] | 0.48 [0.37 to 0.62]
  PnC-IgG-ELISA Type 9V: Pre Booster | 0.18 [0.15 to 0.21] | 0.22 [0.16 to 0.28] | 0.83 [0.60 to 1.14]
  PnC-IgG-ELISA Type 9V: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 9V: Post Booster | 2.44 [2.02 to 2.95] | 3.23 [2.76 to 3.79] | 0.76 [0.59 to 0.97]
  PnC-IgG-ELISA Type 14: 4 weeks post Vac 3 | 4.38 [3.51 to 5.46] | 3.71 [2.67 to 5.16] | 1.18 [0.80 to 1.74]
  PnC-IgG-ELISA Type 14: Pre Booster | 0.81 [0.64 to 1.03] | 1.52 [1.18 to 1.97] | 0.53 [0.38 to 0.76]
  PnC-IgG-ELISA Type 14: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 14: Post Booster | 8.16 [6.19 to 10.77] | 7.60 [5.82 to 9.93] | 1.07 [0.73 to 1.57]
  PnC-IgG-ELISA Type 19A: 4 weeks post Vac 3 | 1.35 [1.05 to 1.74] | 5.12 [3.92 to 6.68] | 0.26 [0.18 to 0.38]
  PnC-IgG-ELISA Type 19A: Pre Booster | 0.29 [0.22 to 0.38] | 0.59 [0.43 to 0.80] | 0.49 [0.33 to 0.74]
  PnC-IgG-ELISA Type 19A: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 19A: Post Booster | 6.72 [4.87 to 9.25] | 15.20 [11.83 to 19.54] | 0.44 [0.29 to 0.66]
  PnC-IgG-ELISA Type 19F: 4 weeks post Vac 3 | 3.70 [3.03 to 4.53] | 4.61 [3.86 to 5.51] | 0.80 [0.61 to 1.05]
  PnC-IgG-ELISA Type 19F: Pre Booster | 0.63 [0.49 to 0.80] | 0.59 [0.45 to 0.75] | 1.07 [0.76 to 1.52]
  PnC-IgG-ELISA Type 19F: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 19F: Post Booster | 7.73 [5.96 to 10.03] | 11.85 [9.41 to 14.92] | 0.65 [0.46 to 0.92]
  PnC-IgG-ELISA Type 23F: 4 weeks post Vac 3 | 1.35 [1.06 to 1.73] | 2.18 [1.67 to 2.87] | 0.62 [0.43 to 0.89]
  PnC-IgG-ELISA Type 23F: Pre Booster | 0.23 [0.17 to 0.30] | 0.17 [0.14 to 0.22] | 1.32 [0.93 to 1.87]
  PnC-IgG-ELISA Type 23F: Post Booster: number analyzed (Participants) | 48 | 47 | 95
  PnC-IgG-ELISA Type 23F: Post Booster | 5.11 [3.93 to 6.65] | 5.28 [4.04 to 6.90] | 0.97 [0.67 to 1.40]

19. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) in Immunoglobulin G (IgG) Among Infants Receiving a Booster Dose
Description: Using enzyme-linked immunosorbent assay (ELISA). Blood samples were collected for immunogenicity testing before and 28 days after the booster dose for infants.
Time Frame: 4 weeks (28 days)
Population: This population is infants who had a booster vaccination of either PCV-10 or Prevenar-13. The evaluable group differs for individual serotypes due to NR results.
Measure: Geometric Mean (90% Confidence Interval); unit: fold change
Groups:
- GMFR Ratio: This column is the GMFR ratio between the SIILPCV 10 group and the Prevenar 13 group.
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13 | GMFR Ratio
Number analyzed (Participants) | 48 | 47 | 95
fold change
  PnC-IgG-ELISA type 1 | 22.52 [17.60 to 28.82] | 15.75 [12.16 to 20.41] | 1.43 [1.00 to 2.04]
  PnC-IgG-ELISA type 5 | 14.83 [12.32 to 17.85] | 10.17 [8.62 to 11.99] | 1.46 [1.14 to 1.86]
  PnC-IgG-ELISA type 6A: number analyzed (Participants) | 48 | 46 | 94
  PnC-IgG-ELISA type 6A | 20.70 [16.13 to 26.56] | 22.98 [17.88 to 29.54] | 0.90 [0.63 to 1.28]
  PnC-IgG-ELISA type 6B: number analyzed (Participants) | 48 | 45 | 93
  PnC-IgG-ELISA type 6B | 17.81 [14.55 to 21.80] | 28.66 [23.43 to 35.05] | 0.62 [0.47 to 0.82]
  PnC-IgG-ELISA type 7F | 13.37 [10.86 to 16.45] | 10.44 [8.59 to 12.70] | 1.28 [0.96 to 1.70]
  PnC-IgG-ELISA type 9V | 13.48 [11.26 to 16.13] | 15.02 [11.73 to 19.23] | 0.90 [0.66 to 1.21]
  PnC-IgG-ELISA type 14 | 10.03 [7.38 to 13.63] | 4.99 [3.78 to 6.60] | 2.01 [1.33 to 3.03]
  PnC-IgG-ELISA Type 19A | 23.20 [15.67 to 34.36] | 25.73 [18.25 to 36.28] | 0.90 [0.54 to 1.51]
  PnC-IgG-ELISA Type 19F: number analyzed (Participants) | 48 | 45 | 93
  PnC-IgG-ELISA Type 19F | 12.44 [8.74 to 17.72] | 20.60 [14.68 to 28.92] | 0.60 [0.37 to 0.98]
  PnC-IgG-ELISA Type 23F | 22.10 [17.30 to 28.23] | 30.75 [23.34 to 40.52] | 0.72 [0.50 to 1.03]

20. Other Pre Specified Outcome: Antibody Persistence of Immunoglobulin G (IgG) Geometric Mean Concentration Among Infants Receiving a Booster Dose
Description: Defined as the ratio of IgG geometric mean concentration (GMC) measured prior to the infant booster dose, to GMC measured 4 weeks after the 3-dose primary series. Infants received the booster dose at least four weeks after they received routine Expanded Program on Immunization (EPI) vaccines, which occurred at 9 months of age. Thus, the time frame was at least 20 weeks but may have been longer.
Time Frame: 20-23 weeks
Population: This population is infants who had a booster vaccination of either PCV-10 or Prevenar-13. The evaluable group differs for individual serotypes due to non-reportable results.
Measure: Geometric Mean (90% Confidence Interval); unit: concentration ratio
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 49 | 47
concentration ratio
  PnC-IgG-ELISA type 1 | 0.10 [0.08 to 0.13] | 0.10 [0.08 to 0.13]
  PnC-IgG-ELISA type 5 | 0.08 [0.06 to 0.10] | 0.17 [0.13 to 0.23]
  PnC-IgG-ELISA type 6A | 0.43 [0.30 to 0.61] | 0.34 [0.24 to 0.49]
  PnC-IgG-ELISA type 6B | 0.52 [0.36 to 0.75] | 0.14 [0.10 to 0.19]
  PnC-IgG-ELISA type 7F | 0.25 [0.18 to 0.34] | 0.24 [0.18 to 0.31]
  PnC-IgG-ELISA type 9V | 0.17 [0.13 to 0.22] | 0.10 [0.07 to 0.13]
  PnC-IgG-ELISA type 14 | 0.19 [0.13 to 0.26] | 0.41 [0.27 to 0.62]
  PnC-IgG-ELISA Type 19A | 0.22 [0.15 to 0.31] | 0.12 [0.08 to 0.17]
  PnC-IgG-ELISA Type 19F | 0.17 [0.12 to 0.23] | 0.13 [0.09 to 0.17]
  PnC-IgG-ELISA Type 23F | 0.17 [0.12 to 0.24] | 0.08 [0.06 to 0.11]

21. Other Pre Specified Outcome: Booster Effect: Ratio of Immunoglobulin G (IgG) Geometric Mean Concentration 4 Weeks Post Vaccination 3 Versus 4 Weeks Post Booster Among Infants Receiving a Booster Dose
Description: Defined as the ratio of IgG geometric mean concentration (GMC) measured 4 weeks post-infant booster dose, to GMC measured 4 weeks after the 3-dose primary series. Infants received the booster dose at least four weeks after they received routine Expanded Program on Immunization (EPI) vaccines, which occurred at 9 months of age. Thus, the time frame was at least 24 weeks but may have been longer.
Time Frame: 24-26 weeks
Population: as for outcome 20
Measure: Geometric Mean (90% Confidence Interval); unit: concentration ratio
Arm/Group | Infant--PCV 10 | Infant--Prevenar 13
Number analyzed (Participants) | 49 | 47
concentration ratio
  PnC-IgG-ELISA type 1 | 2.34 [1.65 to 3.31] | 1.58 [1.17 to 2.13]
  PnC-IgG-ELISA type 5 | 1.14 [0.88 to 1.48] | 1.77 [1.33 to 2.35]
  PnC-IgG-ELISA type 6A | 8.93 [5.86 to 13.62] | 7.75 [5.53 to 10.85]
  PnC-IgG-ELISA type 6B | 9.18 [6.18 to 13.63] | 3.83 [2.70 to 5.43]
  PnC-IgG-ELISA type 7F | 3.40 [2.51 to 4.59] | 2.48 [1.89 to 3.25]
  PnC-IgG-ELISA type 9V | 2.31 [1.79 to 2.98] | 1.46 [1.14 to 1.86]
  PnC-IgG-ELISA type 14 | 1.87 [1.31 to 2.65] | 2.05 [1.35 to 3.12]
  PnC-IgG-ELISA Type 19A | 4.96 [3.32 to 7.41] | 2.97 [2.07 to 4.27]
  PnC-IgG-ELISA Type 19F | 2.09 [1.51 to 2.89] | 2.57 [1.93 to 3.42]
  PnC-IgG-ELISA Type 23F | 3.78 [2.65 to 5.40] | 2.42 [1.66 to 3.52]

ADVERSE EVENTS:
Time Frame: All adult and toddler subjects were monitored for AEs until 28 days after receipt of vaccine, and ongoing AEs at study exit were followed until last subject last visit (LSLV). Infant subjects were monitored for AEs until 28 days after receipt of three doses of the vaccine. For infants who participated in the booster phase of the study, AEs were recorded at 28 days post booster dose, and any conditions present at the visit when booster dose was given were considered baseline.
Groups:
- Adult SIILPCV 10; Toddler SIILPCV 10: Single dose of SIILPCV10 on Day 0
- Infants SIILPCV 10: A 3-dose series of SIILPCV 10 on Days 0, 28, & 56
- Infants Prevenar 13: A 3-dose series of Prevenar 13 on Days 0, 28, & 56
- Booster Infants SIILPCV 10: Booster dose of SIILPCV 10 at 9 months of age
- Booster Infants Prevenar 13: Booster dose of Prevenar 13 at 9 months of age
Arm/Group | Adult SIILPCV 10 | Adult Pneumovax 23 | Toddler SIILPCV 10 | Toddler Prevenar 13 | Infants SIILPCV 10 | Infants Prevenar 13 | Booster Infants SIILPCV 10 | Booster Infants Prevenar 13
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/56 | 0/56 | 0/100 | 0/100 | 0/49 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 1/56 | 1/56 | 6/100 | 2/100 | 1/49 | 0/47
Other Adverse Events (participants affected / at risk) | 4/17 | 10/17 | 35/56 | 36/56 | 97/100 | 96/100 | 25/49 | 24/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult SIILPCV 10 (N=17) | Adult Pneumovax 23 (N=17) | Toddler SIILPCV 10 (N=56) | Toddler Prevenar 13 (N=56) | Infants SIILPCV 10 (N=100) | Infants Prevenar 13 (N=100) | Booster Infants SIILPCV 10 (N=49) | Booster Infants Prevenar 13 (N=47)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult SIILPCV 10 (N=17) | Adult Pneumovax 23 (N=17) | Toddler SIILPCV 10 (N=56) | Toddler Prevenar 13 (N=56) | Infants SIILPCV 10 (N=100) | Infants Prevenar 13 (N=100) | Booster Infants SIILPCV 10 (N=49) | Booster Infants Prevenar 13 (N=47)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (7) | 5 (6) | 29 (34) | 22 (22) | 2 (2) | 5 (5)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pruritis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 55 (72) | 61 (77) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 8 (8) | 9 (9) | 64 (90) | 48 (72) | 14 (16) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 9 (9) | 3 (3) | 1 (1) | 3 (3)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Rash Pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (4)
Vaccination site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 4 (4) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 6 (6) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 27 (29) | 19 (20) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 8 (8) | 6 (7) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 5 (5) | 19 (20) | 17 (21) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 8 (8) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 31 (35) | 21 (24) | 0 (0) | 0 (0)
Cough (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 7 (7) | 0 (0) | 0 (0)
Papular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 8 (9) | 0 (0) | 0 (0)
Microcytic anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No